CLINICAL TRIAL: NCT02125240
Title: Icotinib as an Adjuvant Therapy for Stage II-IIIA Adenocarcinoma With EGFR Mutation: A Placebo-controlled, Randomized, Double-blind, Phase III Study
Brief Title: Icotinib Versus Placebo as Adjuvant Therapy in EGFR-mutant Lung Adenocarcinoma
Acronym: ICWIP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BD-IC-IV-59
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer; Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — icotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Icotinib (Experimental): 125 mg three times daily (375 mg per day) by mouth
  Interventions: Drug: Icotinib
- Placebo (Active Comparator): 1 tablet three times daily by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Icotinib — 125 mg three times daily (375 mg per day) by mouth
  Other Names: BPI-2009; Conmana
  Arms: Icotinib
Drug: Placebo — 1 tablet three times daily by mouth
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare 3years of disease-free survival (DFS) of Icotinib and placebo in the treatment of patients who EGFR mutation-positive II-IIIA lung adenocarcinoma.

DETAILED DESCRIPTION:
This study is designed to compare 3 years of disease-free survival (DFS) of Icotinib and placebo in the treatment of patients who EGFR mutation-positive II-IIIA lung adenocarcinoma.

Primary Outcome Measure:

Disease-free survival between Icotinib group and placebo group.

Secondary Outcome Measures:

Overall survival between Icotinib group and placebo group. Lung cancer symptoms and health-related quality of life (HRQoL) . Number of participants with adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed lung adenocarcinoma after surgical resection
* Stage II-IIIA disease according to 7th edition of TNM staging
* Patients must harbor sensitive EGFR gene mutation (19/21)
* Received four cycles of platinum-based adjuvant chemotherapy.There are many different kinds of chemotherapy regimens including vinorelbine, gemcitabine, docetaxel, paclitaxel, pemetrexed plus cisplatin or carboplatin.The first cycle of chemotherapy with cisplatin dose of 75 mg / m2 ± 10% or carboplatin AUC = 5 ± 10% to calculate the dose of chemotherapy

Exclusion Criteria:

* Previous systemic anti-tumor therapy, including chemotherapy or targeted therapy(Including but not limited to monoclonal antibodies, small molecule tyrosine kinase inhibitor, etc
* Presence of metastatic disease
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Any unresolved chronic toxicity from previous anticancer therapy
* Received antitumor radiation therapy (except for the stage IIIA N2 patients who received adjuvant radiotherapy after surgery)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-12 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 36 months
  DFS was defined as the time from the date of first dose of study medication to the date of death due to disease recurrence or disease progression.

SECONDARY OUTCOMES:
Overall survival | 60 months
  OS was assessed via calculation of the time to death due to any cause from the date of randomization. A patient was censored at the last date they were known to be alive.
Lung cancer symptoms and health-related quality of life (HRQoL) differences | 60 months
Number of participants with adverse events | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Kai Shi, MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (11):
- China (11):
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - China-japan friendship hospital in Beijing, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - 304 Hospital of PLA, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - People's Liberation Army General Hospital (301 Hospital), Beijing, Beijing Municipality
  - Capital Medical University, Beijing Chest Hospital, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Liu YT, Hao XZ, Liu DR, Cheng G, Zhang SC, Xiao WH, Hu Y, Liu JF, He M, Ding CM, Zhang L, Wang J, Li H, Dong GL, Zhi XY, Li J, Shi YK. Icotinib as Adjuvant Treatment for Stage II-IIIA Lung Adenocarcinoma Patients with EGFR Mutation (ICWIP Study): Study Protocol for a Randomised Controlled Trial. Cancer Manag Res. 2020 Jun 17;12:4633-4643. doi: 10.2147/CMAR.S240275. eCollection 2020. PMID 32606956